CLINICAL TRIAL: NCT00792428
Title: Facilitating Motor Recovery After Stroke Using tDCS
Brief Title: Non-invasive Brain Stimulation and Occupational Therapy To Enhance Stroke Recovery
Acronym: TDCS+OT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gottfried Schlaug, Associate Professor of Neurology; Staff Neurologist, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005P000346; R01NS045049 (NIH)
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Cerebrovascular Accident; CVA; Acute Stroke; Acute Cerebrovascular Accident; Apoplexy
Keywords: Stroke; Ischemia; Infarction; Cerebrovascular Disorder; Central Nervous System Diseases; Brain Infarction; Brain Ischemia; Rehabilitation; Recovery; Neurorehabilitation; Plasticity
MeSH Terms: conditions — Stroke; Ischemia; Infarction; Cerebrovascular Disorders; Central Nervous System Diseases; Brain Infarction; Brain Ischemia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real-tDCS + PT-OT (Active Comparator): Each subject will receive up to 5 days of traditional physical-occupational therapy for at least 1 hour per day in the stroke recovery laboratory in combination with real transcranial direct current stimulation (tDCS) over the motor region for up to 30 min.
  Interventions: Device: Real Transcranial Direct Current Stimulation
- Sham-tDCS + PT-OT (Sham Comparator): Each subject will receive up to 5 days of traditional physical-occupational therapy for at least 1 hour per day in the stroke recovery laboratory in combination with sham (pretend) tDCS for up to 30 min. over the motor region.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Real Transcranial Direct Current Stimulation — A direct current runs between two electrode positions and affects the excitability of the underlying brain tissue
  Other Names: Non-invasive brain stimulation; Brain stimulation; Enhancing stroke recovery
  Arms: Real-tDCS + PT-OT
Device: Sham Transcranial Direct Current Stimulation — A sham current runs between two electrode positions and might affect the underlying brain tissue.
  Other Names: Non-invasive brain stimulation; Brain stimulation; Enhancing stroke recovery
  Arms: Sham-tDCS + PT-OT

SUMMARY:
The purpose of this study is to determine whether a non-painful, non-invasive, brain-stimulation technique called transcranial direct current stimulation (tDCS) combined with traditional physical-occupational therapy (OT) will improve motor function in patients with chronic stroke. The aim is to determine the effect of applying real (anodal and/or cathodal) - in a dual configuration - vs sham (pretend) tDCS to the motor brain regions on both hemispheres - in a dual configuration - to improve motor function in chronic stroke patients. Our research in normal subjects has shown that motor skills can be enhanced if tDCS is applied to the brain's motor region during motor learning. The effects after a single session of tDCS can last for up to 30 minutes, effects of multiple sessions (one session per day) can last for weeks. Furthermore, single sessions of tDCS applied to the motor regions in stroke patients have shown that improvements in motor functions can be seen and that effects may last for at least 30 minutes. Patients enrolled in this trial will be randomized to receive either real tDCS or sham tDCS in combination with PT-OT once a day for 5 days. Assessments will be done about 3 days and 7 days after the end of the experimental treatment by investigators who are blinded to the intervention. Patients are also blinded as to whether they are receiving real or sham tDCS. We hypothesize that real tDCS applied to the motor regions in combination with PT-OT results in a subsequent improvement in motor function of the recovering hand over sham tDCS in combination with PT-OT.

ELIGIBILITY:
Inclusion Criteria:

* First time clinical ischemic stroke or cerebrovascular accident
* At least 5 months out from first ischemic stroke prior to study enrollment

Exclusion Criteria:

* More than 1 stroke (older strokes)
* Significant pre-stroke disability
* A terminal medical illness or disorder with survival of less than 1 year
* Co-existent major neurological or psychiatric diseases (e.g., epilepsy)
* Use of psychoactive drugs/medications - such as antidepressants,antipsychotic, stimulating agents
* Active participation in other stroke recovery trials testing interventions

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06; Primary Completion 2013-02-01 (Actual); Study Completion 2013-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Schlaug, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center / Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center / Harvard Medical School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vines BW, Nair D, Schlaug G. Modulating activity in the motor cortex affects performance for the two hands differently depending upon which hemisphere is stimulated. Eur J Neurosci. 2008 Oct;28(8):1667-73. doi: 10.1111/j.1460-9568.2008.06459.x. PMID 18973584
- [Background] Vines BW, Cerruti C, Schlaug G. Dual-hemisphere tDCS facilitates greater improvements for healthy subjects' non-dominant hand compared to uni-hemisphere stimulation. BMC Neurosci. 2008 Oct 28;9:103. doi: 10.1186/1471-2202-9-103. PMID 18957075
- [Background] Nair DG, Hutchinson S, Fregni F, Alexander M, Pascual-Leone A, Schlaug G. Imaging correlates of motor recovery from cerebral infarction and their physiological significance in well-recovered patients. Neuroimage. 2007 Jan 1;34(1):253-63. doi: 10.1016/j.neuroimage.2006.09.010. Epub 2006 Oct 27. PMID 17070707
- [Background] Vines BW, Nair DG, Schlaug G. Contralateral and ipsilateral motor effects after transcranial direct current stimulation. Neuroreport. 2006 Apr 24;17(6):671-4. doi: 10.1097/00001756-200604240-00023. PMID 16603933
- [Result] Lindenberg R, Renga V, Zhu LL, Nair D, Schlaug G. Bihemispheric brain stimulation facilitates motor recovery in chronic stroke patients. Neurology. 2010 Dec 14;75(24):2176-84. doi: 10.1212/WNL.0b013e318202013a. Epub 2010 Nov 10. PMID 21068427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We advertised in local media, on Craig's list, and informed neurology colleagues and rehabilitation specialists about our trial. Stroke patients had to be at least 5 months out from their stroke and had to have a moderate impairment in their upper extremity weakness.
Pre-assignment Details: There were no significant events that occurred after participant enrollment, prior to assignment.
Period: Overall Study
Arm/Group | Real-tDCS + PT-OT | Sham-tDCS + PT-OT
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real-tDCS + PT-OT | Sham-tDCS + PT-OT | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (14.7) | 55.8 (12.9) | 58.7 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment of Upper Extremity Motor Impairment
Description: This scale goes from 0 to 66 (max). Higher values are considered to be a better outcome.
Time Frame: Baseline Assessment; 3 days after 5 treatment days; 7 days after 5 treatment days
Measure: Mean (Standard Deviation); unit: units on a scale [0-66]
Groups:
- Real-tDCS + PT-OT: Subjects are receiving real tDCS in a dual configuration centered over the motor region on both hemispheres for 30 minutes while they are also receiving PT-OT for 60 minutes total.
- Sham-tDCS + PT-OT: Subjects are receiving sham tDCS in a dual configuration centered over the motor region on both hemispheres for 30 minutes while they are also receiving PT-OT for 60 minutes total.
Arm/Group | Real-tDCS + PT-OT | Sham-tDCS + PT-OT
Number analyzed (Participants) | 10 | 10
units on a scale [0-66]
  Pre-treatment (Baseline) | 38.2 (13.3) | 39.8 (11.5)
  Post-treatment1 (3 days after 5 days of treatment) | 43.8 (12.3) | 41.0 (11.8)
  Post-treatment2 (7 days after 5 days of treatment) | 44.3 (11.5) | 40.9 (11.7)

2. Secondary Outcome: Wolf-Motor-Function-Test
Description: The Wolf-Motor-Function-Test (time) is the average time in seconds taken to perform each of 15 functional tasks ranging in difficulty from putting one's forearm on a table to stacking checkers. Participants are given 120 seconds to perform a task and if they fail, they are scored 120 for that task," or similar as accurate. The average time in seconds is then log10 transformed.
Time Frame: Baseline Assessment; 3 days after 5 treatment days; 7 days after 5 treatment days
Measure: Mean (Standard Deviation); unit: units on a scale (log(sec))
Arm/Group | Real-tDCS + PT-OT | Sham-tDCS + PT-OT
Number analyzed (Participants) | 10 | 10
units on a scale (log(sec))
  Pre-treatment (baseline) | 0.87 (0.55) | 0.83 (0.48)
  Post-treatment1 (3 days after 5 days of treatment) | 0.74 (0.49) | 0.79 (0.47)
  Post-treatment2 (7 days after 5 days of treatment) | 0.73 (0.49) | 0.78 (0.46)

ADVERSE EVENTS:
Time Frame: Over the 5 days of experimental treatment and during the 1 week follow-up.
Groups:
- Sham tDCS + PT-OT: Subjects are receiving sham tDCS in a dual configuration over both motor regions for 30 minutes while they are also receiving PT-OT for 60 minutes
Arm/Group | Real-tDCS + PT-OT | Sham tDCS + PT-OT
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No